CLINICAL TRIAL: NCT01814826
Title: A Phase 1b, Open-Label, Dose-Escalation Study of MLN4924 Plus Azacitidine in Treatment-Naïve Patients With Acute Myelogenous Leukemia Who Are 60 Years or Older
Brief Title: Study of MLN4924 Plus Azacitidine in Treatment-naive Participants With Acute Myelogenous Leukemia (AML) Who Are 60 Years or Older
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: C15009; U1111-1221-2792 (Other: WHO)
Record Dates: First submitted 2013-03-18; First posted 2013-03-20 (Estimated); Results first posted 2020-03-03 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Acute Myelogenous Leukemia
Keywords: Drug Therapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — pevonedistat; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MLN4924 and Azacitidine (Experimental)
  Interventions: Drug: MLN4924; Drug: Azacitidine

INTERVENTIONS:
Drug: MLN4924 — MLN4924 intravenously (IV) in AML participants in a 28-day cycle:
  * MLN4924 on Days 1, 3, and 5 for Cycle 1 and all subsequent cycles
  Other Names: Pevonedistat
Drug: Azacitidine — Azacitidine (IV) or subcutaneously in AML participants in a 28-day cycle:
  - Azacitidine Days 1, 2, 3, 4, 5, 8, 9 in Cycle 1 and for all subsequent cycles

SUMMARY:
The purpose of this study is to establish the maximum tolerated dose (MTD), and to assess the safety and tolerability of MLN4924 (pevonedistat) in combination with azacitidine in treatment naive participants with AML who were 60 years of age or older.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with world health organization (WHO)-defined AML, 60 years of age or older, who are unlikely to benefit from standard induction therapy, defined as having at least 1 of the following:

   * Greater than or equal to 75 years of age.
   * Antecedent hematologic disease.
   * Known adverse cytogenetic risk.
   * Eastern Cooperative Oncology Group (ECOG) PS = 2.
   * Participant must not have received definitive treatment for AML, defined as any prior chemotherapy with antileukemic activity.
2. ECOG PS 0 to 2.
3. Expected survival longer than 3 months from enrollment in the study.
4. Female participants who are post menopausal, surgically sterile, or agree to practice 2 effective methods of contraception or agree to practice true abstinence.
5. Male participants who agree to practice effective barrier contraception or agree to practice true abstinence.
6. Voluntary written consent must be given before performance of any study-related procedure.
7. Suitable venous access for the study-required blood sampling.
8. Clinical laboratory values as specified below within 3 days before the first dose of any study drug:

   •Total bilirubin must be less than or equal to (<=) the upper limit of the normal range (ULN).
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) must be<=2.5*ULN.
   * Serum creatinine <=1.5*ULN.
   * Albumin greater than or equal to (>=) 27 grams per liter (g/L).
   * Hemoglobin >9 grams per deciliter (g/dL). Note: It was permissible to transfuse participants with red blood cells to achieve this criterion.
   * White blood cell (WBC) count less than (<) 50,000 per microliter (/mcL) before administration of pevonedistat on Days 1, 3, and 5 of Cycle 1.

   Note: Hydroxyurea could be used to control the level of circulating leukemic blast cell counts to no lower than 10,000/mcL while on pevonedistat.
9. Able to undergo bone marrow aspiration and biopsy at screening.

Exclusion Criteria:

1. Previous treatment with azacitidine or decitabine.
2. Known favorable cytogenetic risk.
3. Any serious medical or psychiatric illness.
4. Treatment with any investigational products.
5. Known hypersensitivity to azacitidine or mannitol.
6. Acute promyelocytic leukemia as diagnosed by morphologic examination of bone marrow, by fluorescent in situ hybridization or cytogenetics of peripheral blood or bone marrow, or by other accepted analysis.
7. Active uncontrolled infection or severe infectious disease.
8. Major surgery within 14 days before the first dose of study drug.
9. Life-threatening illness unrelated to cancer.
10. Clinically uncontrolled central nervous system (CNS) involvement.
11. WBC count greater than (>) 50,000/ mcL.
12. Prothrombin time (PT) or activated partial thromboplastin time (aPTT) >1.5* ULN or a history of coagulopathy or bleeding disorder
13. Known human immunodeficiency virus (HIV) positive.
14. Known hepatitis B surface antigen-positive, or known or suspected active hepatitis C infection
15. Known hepatic cirrhosis or severe pre-existing hepatic impairment.
16. Known cardiac/cardiopulmonary disease defined as 1 of the following:

    * Uncontrolled high blood pressure (that is, systolic blood pressure >180 milliliter per mercury (mm Hg), diastolic blood pressure >95 mm Hg).
    * Congestive heart failure New York Heart Association (NYHA) Class III or IV, or Class II with a recent decompensation that required hospitalization or referral to a heart failure clinic within 4 weeks before screening (see Section 15.4 of the protocol in Appendix 16.1.1).
    * Cardiomyopathy or history of ischemic heart disease
    * Participants with ischemic heart disease who had acute coronary syndrome (ACS), myocardial infarction (MI), and/or revascularization (example, coronary artery bypass graft, stent) in the past 6 months were excluded. However, participants with ischemic heart disease who had ACS, MI, and/or revascularization greater than 6 months before screening and who are without cardiac symptoms could be enrolled.
    * Arrhythmia (example, history of polymorphic ventricular fibrillation or torsade de pointes). However, participants with <Grade 3 atrial fibrillation (a fib) for a period of at least 6 months could enroll. Grade 3 a fib is symptomatic and incompletely controlled medically, or controlled with device (example, pacemaker), or ablation. Participants with paroxysmal a fib were permitted to enroll.
    * Implantable cardioverter defibrillator.
    * Moderate to severe aortic and/or mitral stenosis or other valvulopathy (ongoing).
    * Pulmonary arterial hypertension. Prolonged rate corrected QT (QTc) interval >= 500 msec, calculated according to institutional guidelines
17. Left ventricular ejection fraction
18. Known moderate to severe chronic obstructive pulmonary disease, interstitial lung disease, and pulmonary fibrosis.
19. Body mass index >40 kilogram per square meter (kg/m^2).
20. Treatment with CYP3A inducers within 14 days before the first dose of MLN4924.
21. Systemic antineoplastic therapy or radiotherapy within 14 days before the first dose of study drug, except for hydroxyurea.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2013-04-10 (Actual); Primary Completion 2016-05-03 (Actual); Study Completion 2018-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (8):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University, Stanford, California
  - Hospital Corporation of America-HealthOne, LLC, Denver, Colorado
  - Mayo Clinic - Jacksonville, FL, Jacksonville, Florida
  - University of Miami School of Medicine, Miami, Florida
  - UNC-Chapel Hill School of Medicine, Chapel Hill, North Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Methodist Hospital, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Result] Swords RT, Coutre S, Maris MB, Zeidner JF, Foran JM, Cruz J, Erba HP, Berdeja JG, Tam W, Vardhanabhuti S, Pawlikowska-Dobler I, Faessel HM, Dash AB, Sedarati F, Dezube BJ, Faller DV, Savona MR. Pevonedistat, a first-in-class NEDD8-activating enzyme inhibitor, combined with azacitidine in patients with AML. Blood. 2018 Mar 29;131(13):1415-1424. doi: 10.1182/blood-2017-09-805895. Epub 2018 Jan 18. PMID 29348128
- [Derived] Faessel HM, Mould DR, Zhou X, Faller DV, Sedarati F, Venkatakrishnan K. Population pharmacokinetics of pevonedistat alone or in combination with standard of care in patients with solid tumours or haematological malignancies. Br J Clin Pharmacol. 2019 Nov;85(11):2568-2579. doi: 10.1111/bcp.14078. Epub 2019 Sep 4. PMID 31355467

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 8 investigative sites in the United states from 10 April 2013 to 08 April 2018.
Pre-assignment Details: Participants diagnosed with acute myelogenous leukemia (AML) were enrolled to receive MLN4924 in combination with azacitidine intravenous during dose-escalation phase and MLN4924 in combination with azacitidine intravenous or subcutaneous during expansion phase.
Groups:
- MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous: MLN4924 20 mg/m^2, infusion, intravenously, once on Days 1, 3, and 5 in combination with azacitidine 75 mg/m^2, infusion, intravenously, once on Days 1 through 5, 8 and 9 before administration of MLN4924 in a 28-day treatment cycle up to symptomatic deterioration or progressive disease (PD), or until treatment was discontinued for another reason (up to Cycle 53).
- MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Subcutaneous: MLN4924 20 mg/m^2, infusion, intravenously, once on Days 1, 3, and 5 in combination with azacitidine 75 mg/m^2, infusion, subcutaneously, once on Days 1 through 5, 8 and 9 before administration of MLN4924 in a 28-day treatment cycle up to symptomatic deterioration or PD, or until treatment was discontinued for another reason (up to Cycle 53).
- MLN4924 30 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous: MLN4924 30 mg/m^2, infusion, intravenously, once on Days 1, 3, and 5 in combination with azacitidine 75 mg/m^2, infusion, intravenously, once on Days 1 through 5, 8 and 9 before administration of MLN4924 in a 28-day treatment cycle up to symptomatic deterioration or PD, or until treatment was discontinued for another reason (up to Cycle 53).
Period: Overall Study
Arm/Group | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Subcutaneous | MLN4924 30 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous
Started | 32 (6 participants were enrolled into the dose escalation phase and 26 in the MTD expansion phase.) | 29 (29 participants were enrolled into the MTD expansion phase.) | 3 (3 participants were enrolled into the dose escalation phase.)
Completed | 0 | 0 | 0
Not Completed | 32 | 29 | 3
Not completed — Other | 3 | 5 | 0
Not completed — Death | 29 | 24 | 3

BASELINE CHARACTERISTICS:
Population: The safety population was defined as all enrolled participants who receive at least 1 dose of any study drug, MLN4924 or azacitidine.
Groups:
- Total: Total of all reporting groups
Arm/Group | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Subcutaneous | MLN4924 30 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous | Total
Number analyzed (Participants) | 32 | 29 | 3 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.7 (6.28) | 75.2 (6.00) | 80.3 (3.21) | 75.2 (6.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 2 | 30
  Male | 18 | 15 | 1 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 0 | 8
  Not Hispanic or Latino | 28 | 22 | 3 | 53
  Unknown or Not Reported | 1 | 2 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 0 | 0 | 4
  White | 27 | 28 | 3 | 58
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32 | 29 | 3 | 64
Body Surface Area (BSA) [Mean (Standard Deviation); unit: square meter (m^2)] | 1.88 (0.249) | 1.85 (0.256) | 1.79 (0.428) | 1.86 (0.257)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: Baseline up to 30 days after the last dose of study drug (up to 5 years)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Subcutaneous | MLN4924 30 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous
Number analyzed (Participants) | 32 | 29 | 3
Participants
  TEAEs | 32 | 29 | 3
  SAEs | 21 | 22 | 3

2. Primary Outcome: Number of Participants With TEAEs Related to Clinically Significant Laboratory Evaluation Findings
Time Frame: Baseline up to 30 days after the last dose of study drug (up to 5 years)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Subcutaneous | MLN4924 30 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous
Number analyzed (Participants) | 32 | 29 | 3
Participants
  Blood creatinine increased | 6 | 3 | 2
  Proteinuria | 1 | 0 | 0
  Blood urea increased | 1 | 1 | 0
  Renal impairment | 0 | 1 | 0
  Blood bilirubin increased | 3 | 1 | 1
  Aspartate aminotransferase increased | 5 | 2 | 2
  Alanine aminotransferase increased | 6 | 3 | 2
  Gamma-glutamyltransferase increased | 1 | 2 | 1
  Blood alkaline phosphatase increased | 7 | 0 | 2
  Anaemia | 15 | 10 | 1
  Neutropenia | 10 | 6 | 0
  Leukopenia | 5 | 2 | 1
  Febrile neutropenia | 7 | 12 | 1
  Neutrophil count decreased | 6 | 1 | 0

3. Primary Outcome: Number of Participants With TEAEs Related to Clinically Significant Vital Sign Findings
Time Frame: Baseline up to 30 days after the last dose of study drug (up to 5 years)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Subcutaneous | MLN4924 30 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous
Number analyzed (Participants) | 32 | 29 | 3
Participants
  Tachycardia | 4 | 1 | 0
  Hypotension | 3 | 6 | 0
  Orthostatic Hypotension | 1 | 0 | 0

4. Secondary Outcome: Dose-escalation Phase, Cmax: Maximum Observed Plasma Concentration for MLN4924
Time Frame: Cycle 1 Day 1 pre-dose and at multiple time points (up to 24 hours) post-dose; Cycle 1 Day 5 pre-dose and at multiple time points (up to 48 hours) post-dose (Cycle length is equal to [=] 28 days)
Population: The pharmacokinetic (PK)-evaluable population was defined as all enrolled participants who had sufficient dosing in Cycle 1 and MLN4924 concentration-time data to reliably estimate PK parameters. The PK population where data at specified time points was available.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous | MLN4924 30 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous
Number analyzed (Participants) | 6 | 3
nanogram per milliliter (ng/mL)
  Cycle 1 Day 1 | 173.60 (78.017) | 306.67 (81.304)
  Cycle 1 Day 5: number analyzed (Participants) | 6 | 1
  Cycle 1 Day 5 | 177.87 (67.767) | NA (NA) — Mean and Standard deviation could not be evaluated since greater than 50% of the concentration at a given time point were not quantifiable or reportable.

5. Secondary Outcome: Maximum Tolerated Dose (MTD) Expansion Phase, Cmax: Maximum Observed Plasma Concentration for MLN4924
Time Frame: Cycle 1 Day 1 pre-dose and at multiple time points (up to 24 hours) post-dose; Cycle 1 Day 5 pre-dose and at multiple time points (up to 48 hours) post-dose (Cycle length = 28 days)
Population: The PK-evaluable population was defined as all enrolled participants who had sufficient dosing in Cycle 1 and MLN4924 concentration-time data to reliably estimate PK parameters. The PK population where data at specified time points was available.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Subcutaneous
Number analyzed (Participants) | 26 | 28
ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 26 | 27
  Cycle 1 Day 1 | 168.80 (80.504) | 159.78 (57.755)
  Cycle 1 Day 5: number analyzed (Participants) | 18 | 25
  Cycle 1 Day 5 | 176.65 (76.628) | 158.95 (60.807)

6. Secondary Outcome: Dose-escalation Phase, Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for MLN4924
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Median (Full Range); unit: hour
Arm/Group | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous | MLN4924 30 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous
Number analyzed (Participants) | 6 | 3
hour
  Cycle 1 Day 1 | 1.06 [1.0 to 2.3] | 1.0 [1.0 to 1.0]
  Cycle Day 5: number analyzed (Participants) | 6 | 1
  Cycle Day 5 | 1.0 [1.0 to 1.5] | NA [1.0 to 1.0] — Median could not be calculated since only 1 participant was available for analysis.

7. Secondary Outcome: MTD Expansion Phase, Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for MLN4924
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Median (Full Range); unit: hour
Arm/Group | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Subcutaneous
Number analyzed (Participants) | 26 | 28
hour
  Cycle 1 Day 1: number analyzed (Participants) | 26 | 27
  Cycle 1 Day 1 | 1.01 [0.7 to 2.0] | 1.00 [0.9 to 3.0]
  Cycle 1 Day 5: number analyzed (Participants) | 18 | 25
  Cycle 1 Day 5 | 1.0 [0.9 to 2.0] | 0.98 [0.8 to 2.0]

8. Secondary Outcome: Dose-escalation Phase, Ctrough: Observed Plasma Concentration at the End of the Dosing Interval for MLN4924
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous | MLN4924 30 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous
Number analyzed (Participants) | 6 | 3
ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 5 | 3
  Cycle 1 Day 1 | 2.34 (1.987) | 1.68 (0.450)
  Cycle 1 Day 5: number analyzed (Participants) | 6 | 1
  Cycle 1 Day 5 | 1.40 (0.208) | NA (NA) — Mean and Standard deviation could not be evaluated since greater than 50% of the concentration at a given time point were not quantifiable or reportable.

9. Secondary Outcome: MTD Expansion Phase, Ctrough: Observed Plasma Concentration at the End of the Dosing Interval for MLN4924
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Subcutaneous
Number analyzed (Participants) | 26 | 28
ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 23 | 25
  Cycle 1 Day 1 | 0.87 (0.974) | 0.91 (1.105)
  Cycle 1 Day 5: number analyzed (Participants) | 21 | 26
  Cycle 1 Day 5 | 1.51 (1.321) | 1.30 (1.010)

10. Secondary Outcome: Dose-escalation Phase, AUC0-tau: Area Under the Plasma Concentration-time Curve From Time Zero to the End of the Dosing Interval (Tau) for MLN4924
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hour*nanogram per milliliter (hr*ng/mL)
Arm/Group | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous | MLN4924 30 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous
Number analyzed (Participants) | 6 | 3
hour*nanogram per milliliter (hr*ng/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 5 | 3
  Cycle 1 Day 1 | 1151.20 (327.445) | 1805.47 (423.488)
  Cycle 1 Day 5: number analyzed (Participants) | 6 | 1
  Cycle 1 Day 5 | 1139.67 (351.423) | NA (NA) — Mean and Standard deviation could not be evaluated since greater than 50% of the concentration at a given time point were not quantifiable or reportable.

11. Secondary Outcome: MTD Expansion Phase, AUC0-tau: Area Under the Plasma Concentration-time Curve From Time Zero to the End of the Dosing Interval (Tau) for MLN4924
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Subcutaneous
Number analyzed (Participants) | 26 | 28
hr*ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 12 | 11
  Cycle 1 Day 1 | NA (NA) — Mean and standard deviation could not be evaluated since greater than 50% of concentrations at a given time point were not quantifiable or reportable. | NA (NA) — Mean and standard deviation could not be evaluated since greater than 50% of concentrations at a given time point were not quantifiable or reportable.
  Cycle 1 Day 5: number analyzed (Participants) | 13 | 18
  Cycle 1 Day 5 | 1125.90 (276.604) | 1122.91 (244.752)

12. Secondary Outcome: Dose-escalation Phase, AUC24hours: Area Under the Plasma Concentration-time Curve From Time Zero to 24 Hours Post-Dose for MLN4924
Time Frame: Cycle 1 Day 1 pre-dose and at multiple time points (up to 24 hours) post-dose; Cycle 1 Day 5 pre-dose and at multiple time points (up to 24 hours) post-dose (Cycle length = 28 days)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous | MLN4924 30 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous
Number analyzed (Participants) | 6 | 3
hr*ng/mL
  Cycle 1 Day 1 | 1020.32 (267.958) | 1675.41 (398.425)
  Cycle 1 Day 5: number analyzed (Participants) | 6 | 1
  Cycle 1 Day 5 | 1039.54 (342.330) | NA (NA) — Mean and Standard deviation could not be evaluated since greater than 50% of the concentration at a given time point were not quantifiable or reportable.

13. Secondary Outcome: MTD Expansion Phase, AUC24hours: Area Under the Plasma Concentration-time Curve From Time Zero to 24 Hours Post-Dose for MLN4924
Time Frame: as for outcome 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Subcutaneous
Number analyzed (Participants) | 26 | 28
hr*ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 24 | 27
  Cycle 1 Day 1 | 891.89 (261.82) | 926.74 (280.128)
  Cycle 1 Day 5: number analyzed (Participants) | 18 | 24
  Cycle 1 Day 5 | 946.91 (244.081) | 954.07 (240.098)

14. Secondary Outcome: Dose-escalation Phase, AUCinf: Area Under the Plasma Concentration-time Curve Extrapolated to Infinity for MLN4924
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous | MLN4924 30 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous
Number analyzed (Participants) | 6 | 3
hr*ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 5 | 3
  Cycle 1 Day 1 | 1101.81 (310.114) | 1823.68 (420.948)
  Cycle 1 Day 5: number analyzed (Participants) | 0 | 0

15. Secondary Outcome: MTD Expansion Phase, AUCinf: Area Under the Plasma Concentration-time Curve Extrapolated to Infinity for MLN4924
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Subcutaneous
Number analyzed (Participants) | 26 | 28
hr*ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 24 | 27
  Cycle 1 Day 1 | 990.58 (279.282) | 1026.45 (310.47)
  Cycle 1 Day 5: number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Dose-escalation Phase, Lambdaz: Terminal Disposition Phase Rate Constant for MLN4924
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: 1 per hour (1/hr)
Arm/Group | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous | MLN4924 30 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous
Number analyzed (Participants) | 6 | 3
1 per hour (1/hr)
  Cycle 1 Day 1: number analyzed (Participants) | 5 | 3
  Cycle 1 Day 1 | 0.09 (0.013) | 0.09 (0.009)
  Cycle 1 Day 5: number analyzed (Participants) | 6 | 1
  Cycle 1 Day 5 | 0.09 (0.009) | NA (NA) — Mean and Standard deviation could not be evaluated since only one participant was analyzed.

17. Secondary Outcome: MTD Expansion Phase, Lambdaz: Terminal Disposition Phase Rate Constant for MLN4924
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Subcutaneous
Number analyzed (Participants) | 26 | 28
1/hr
  Cycle 1 Day 1: number analyzed (Participants) | 24 | 28
  Cycle 1 Day 1 | 0.10 (0.027) | 0.10 (0.022)
  Cycle 1 Day 5: number analyzed (Participants) | 21 | 25
  Cycle 1 Day 5 | 0.09 (0.028) | 0.09 (0.022)

18. Secondary Outcome: Dose-escalation Phase, t1/2: Terminal Disposition Phase Half-life for MLN4924
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous | MLN4924 30 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous
Number analyzed (Participants) | 6 | 3
hour
  Cycle 1 Day 1: number analyzed (Participants) | 5 | 3
  Cycle 1 Day 1 | 7.80 (1.126) | 7.39 (0.699)
  Cycle 1 Day 5: number analyzed (Participants) | 6 | 1
  Cycle 1 Day 5 | 7.98 (0.818) | NA (NA) — Mean and Standard deviation could not be evaluated since greater than 50% of the concentration at a given time point were not quantifiable or reportable.

19. Secondary Outcome: MTD Expansion Phase, t1/2: Terminal Disposition Phase Half-life for MLN4924
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Subcutaneous
Number analyzed (Participants) | 26 | 28
hour
  Cycle 1 Day 1: number analyzed (Participants) | 24 | 28
  Cycle 1 Day 1 | 7.45 (1.851) | 7.30 (1.762)
  Cycle 1 Day 5: number analyzed (Participants) | 21 | 25
  Cycle 1 Day 5 | 8.07 (2.414) | 7.89 (1.764)

20. Secondary Outcome: Dose-escalation Phase, Rac: Observed Accumulation Ratio for MLN4924
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous | MLN4924 30 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous
Number analyzed (Participants) | 6 | 3
ratio
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0
  Cycle 1 Day 5: number analyzed (Participants) | 5 | 1
  Cycle 1 Day 5 | 0.99 (0.145) | NA (NA) — Mean and Standard deviation could not be evaluated since greater than 50% of the concentration at a given time point were not quantifiable or reportable.

21. Secondary Outcome: MTD Expansion Phase, Rac: Observed Accumulation Ratio for MLN4924
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Subcutaneous
Number analyzed (Participants) | 26 | 28
ratio
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0
  Cycle 1 Day 5: number analyzed (Participants) | 8 | 11
  Cycle 1 Day 5 | NA (NA) — Mean and standard deviation could not be evaluated since greater than 50% of concentrations at a given time point were not quantifiable or reportable. | NA (NA) — Mean and standard deviation could not be evaluated since greater than 50% of concentrations at a given time point were not quantifiable or reportable.

22. Secondary Outcome: Dose-escalation Phase, CLp: Systemic Clearance for MLN4924
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: liter per hour (L/hr)
Arm/Group | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous | MLN4924 30 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous
Number analyzed (Participants) | 6 | 3
liter per hour (L/hr)
  Cycle 1 Day 1: number analyzed (Participants) | 5 | 3
  Cycle 1 Day 1 | 35.69 (10.318) | 29.78 (7.511)
  Cycle 1 Day 5: number analyzed (Participants) | 6 | 1
  Cycle 1 Day 5 | 35.27 (13.701) | NA (NA) — Mean and Standard deviation could not be evaluated since greater than 50% of the concentration at a given time point were not quantifiable or reportable.

23. Secondary Outcome: MTD Expansion Phase, CLp: Systemic Clearance for MLN4924
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Subcutaneous
Number analyzed (Participants) | 26 | 28
L/hr
  Cycle 1 Day 1: number analyzed (Participants) | 24 | 27
  Cycle 1 Day 1 | 41.35 (13.924) | 39.20 (14.191)
  Cycle 1 Day 5: number analyzed (Participants) | 13 | 18
  Cycle 1 Day 5 | 38.10 (12.407) | 34.02 (10.010)

24. Secondary Outcome: Dose-escalation Phase, Vss: Volume of Distribution at Steady-state for MLN4924
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: liter (L)
Arm/Group | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous | MLN4924 30 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous
Number analyzed (Participants) | 6 | 3
liter (L)
  Cycle 1 Day 1: number analyzed (Participants) | 5 | 3
  Cycle 1 Day 1 | 352.06 (148.987) | 257.32 (88.354)
  Cycle 1 Day 5: number analyzed (Participants) | 6 | 1
  Cycle 1 Day 5 | 351.82 (182.744) | NA (NA) — Mean and Standard deviation could not be evaluated since greater than 50% of the concentration at a given time point were not quantifiable or reportable.

25. Secondary Outcome: MTD Expansion Phase, Vss: Volume of Distribution at Steady-state for MLN4924
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Subcutaneous
Number analyzed (Participants) | 26 | 28
liter
  Cycle 1 Day 1: number analyzed (Participants) | 24 | 27
  Cycle 1 Day 1 | 370.53 (141.396) | 348.66 (128.661)
  Cycle 1 Day 5: number analyzed (Participants) | 13 | 18
  Cycle 1 Day 5 | 401.41 (173.087) | 370.97 (175.097)

26. Secondary Outcome: Best Overall Response Rate
Description: Disease response was based on best overall response as determined by an investigator based on revised recommendations of the International Working Group (IWG) Response Criteria for AML. Best overall response rate was defined as percentage of participants who had complete response (CR), partial response (PR), or CR/remission with incomplete blood count recovery (Cri). CR: free of leukemia-related symptoms, absolute neutrophil count (ANC) greater than (>)1.0*10^9 per liter (/L), platelet count greater than or equal to (>=) 100*10^9/L, normal bone marrow with <5 percent (%) blasts and no Auer rods. CRi: As per CR but with residual thrombocytopenia (platelet count <100*10^9/L) or residual neutropenia (ANC <1.0*10^9/L). PR: >=50% decrease bone marrow blasts to 5 to 25% abnormal cells, or CR with less than or equal to (<=) 5% blasts if Auer rods present.
Time Frame: Cycle(C)1Day(D)22 and at C2 between D20 and 28 and at C4 and beyond C4 after completion of every 3rd C between D15 and 28 up to 30 days after last dose of study drug/before start of subsequent antineoplastic therapy, if that occurred sooner(up to 5 years)
Population: The response-evaluable population was defined as all participants who received at least 1 dose of study drug, had measurable disease at baseline, and had at least 1 post baseline disease assessment. Participants who were evaluable at a particular time point for this outcome measure were included in the assessment.
Measure: Number; unit: percentage of participants
Arm/Group | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Subcutaneous | MLN4924 30 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous
Number analyzed (Participants) | 28 | 24 | 2
percentage of participants
  CR | 43 | 33 | 50
  PR | 14 | 13 | 0
  CRi | 4 | 13 | 0

27. Secondary Outcome: Duration of Response
Description: The duration of response was defined in participants with disease response (CR, CRi, or PR) as the time between the first documentation of response and disease progression. Duration of response was determined by an investigator based on revised recommendations of the IWG Response Criteria for AML. CR: free of leukemia-related symptoms, absolute neutrophil count (ANC) greater than (>)1.0*10^9 per liter (/L), platelet count greater than or equal to (>=) 100*10^9/L, normal bone marrow with <5 percent (%) blasts and no Auer rods. CRi: As per CR but with residual thrombocytopenia (platelet count <100*10^9/L) or residual neutropenia (ANC <1.0*10^9/L). PR: >=50% decrease bone marrow blasts to 5 to 25% abnormal cells, or CR with less than or equal to (<=) 5% blasts if Auer rods present.
Time Frame: From the date of first documented CR, PR or CRi up to the date of first disease progression (Up to 5 years)
Population: as for outcome 26
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Subcutaneous | MLN4924 30 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous
Number analyzed (Participants) | 17 | 13 | 0
months | 9.0 [5.52 to 15.54] | 6.0 [2.00 to 14.16] |

28. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from the first dose of study drug to the date of death. The Kaplan-Meier method was used to estimate overall survival, along with the corresponding 95% confidence interval.
Time Frame: From the first dose of study drug up to date of death (up to 5 years)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Subcutaneous | MLN4924 30 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous
Number analyzed (Participants) | 32 | 29 | 3
months | 12.25 [4.53 to 17.12] | 4.93 [3.22 to 14.42] | 5.22 [3.38 to 10.71]

29. Secondary Outcome: Thirty-day Mortality Rate
Time Frame: 30 days after the first dose of study drug in Cycle 1 (Cycle Length=28 days)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Subcutaneous | MLN4924 30 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous
Number analyzed (Participants) | 32 | 29 | 3
percentage of participants | 5 | 6 | 0

30. Secondary Outcome: Sixty-day Mortality Rate
Time Frame: 60 days after the first dose of study drug on Cycle 1 (Cycle Length=28 days)
Population: No participant was analyzed since this outcome measure was not planned to be assessed but added in the protocol summary by error.
Arm/Group | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Subcutaneous | MLN4924 30 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) are adverse events that started after the first dose of study drug and no more than 30 days after the last dose of study drug (up to 5 years)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Subcutaneous | MLN4924 30 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous
All-Cause Mortality (participants affected / at risk) | 29/32 | 24/29 | 3/3
Serious Adverse Events (participants affected / at risk) | 21/32 | 22/29 | 3/3
Other Adverse Events (participants affected / at risk) | 32/32 | 29/29 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous (N=32) | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Subcutaneous (N=29) | MLN4924 30 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous (N=3)
Pneumonia (Infections and infestations) | 3 | 4 | 2
Sepsis (Infections and infestations) | 1 | 2 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 2 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 0
Gingivitis (Infections and infestations) | 1 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0
Pneumonia legionella (Infections and infestations) | 1 | 0 | 0
Pseudomonal bacteraemia (Infections and infestations) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 7 | 9 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 3 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 0
Death (General disorders) | 0 | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 2 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0
Electrocardiogram T wave inversion (Investigations) | 0 | 1 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 2 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0
Embolism (Vascular disorders) | 2 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous (N=32) | MLN4924 20 mg/m^2 + Azacitidine 75 mg/m^2 Subcutaneous (N=29) | MLN4924 30 mg/m^2 + Azacitidine 75 mg/m^2 Intravenous (N=3)
Anaemia (Blood and lymphatic system disorders) | 14 | 10 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 10 | 8 | 2
Neutropenia (Blood and lymphatic system disorders) | 10 | 6 | 0
Leukopenia (Blood and lymphatic system disorders) | 5 | 2 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 4 | 1
Lymphopenia (Blood and lymphatic system disorders) | 2 | 2 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2 | 0
Tachycardia (Cardiac disorders) | 4 | 1 | 0
Palpitations (Cardiac disorders) | 2 | 0 | 0
Dry eye (Eye disorders) | 3 | 1 | 0
Constipation (Gastrointestinal disorders) | 18 | 12 | 1
Nausea (Gastrointestinal disorders) | 15 | 11 | 1
Diarrhoea (Gastrointestinal disorders) | 6 | 9 | 0
Vomiting (Gastrointestinal disorders) | 6 | 9 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 3 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 4 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 2 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 2 | 0
Flatulence (Gastrointestinal disorders) | 0 | 2 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 2 | 0
Oesophageal pain (Gastrointestinal disorders) | 0 | 2 | 0
Fatigue (General disorders) | 16 | 10 | 1
Pyrexia (General disorders) | 9 | 5 | 0
Oedema peripheral (General disorders) | 5 | 5 | 1
Chills (General disorders) | 3 | 6 | 0
Asthenia (General disorders) | 3 | 2 | 0
Injection site erythema (General disorders) | 0 | 5 | 0
Injection site pain (General disorders) | 0 | 5 | 0
Pain (General disorders) | 3 | 2 | 0
Injection site rash (General disorders) | 0 | 3 | 0
Peripheral swelling (General disorders) | 3 | 0 | 0
Gait disturbance (General disorders) | 2 | 0 | 0
Ill-defined disorder (General disorders) | 0 | 2 | 0
Injection site reaction (General disorders) | 0 | 2 | 0
Non-cardiac chest pain (General disorders) | 2 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 3 | 0
Urinary tract infection (Infections and infestations) | 4 | 2 | 0
Sinusitis (Infections and infestations) | 3 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 3 | 0
Rhinovirus infection (Infections and infestations) | 1 | 2 | 0
Folliculitis (Infections and infestations) | 2 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 7 | 3 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 2 | 2 | 0
Laceration (Injury, poisoning and procedural complications) | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 6 | 3 | 2
Blood creatinine increased (Investigations) | 6 | 3 | 1
Weight decreased (Investigations) | 4 | 4 | 0
Aspartate aminotransferase increased (Investigations) | 5 | 2 | 2
Blood alkaline phosphatase increased (Investigations) | 7 | 0 | 2
Neutrophil count decreased (Investigations) | 6 | 1 | 0
Platelet count decreased (Investigations) | 5 | 2 | 0
White blood cell count decreased (Investigations) | 3 | 2 | 0
Blood bilirubin increased (Investigations) | 3 | 1 | 1
Lymphocyte count decreased (Investigations) | 2 | 2 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 2 | 1
White blood cell count increased (Investigations) | 1 | 2 | 0
Activated partial thromboplastin time prolonged (Investigations) | 2 | 0 | 0
Fibrin D dimer increased (Investigations) | 2 | 0 | 0
Lymphocyte count increased (Investigations) | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 10 | 8 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8 | 3 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 8 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 1
Fluid overload (Metabolism and nutrition disorders) | 3 | 1 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 3 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 5 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 6 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Dizziness (Nervous system disorders) | 6 | 4 | 0
Headache (Nervous system disorders) | 4 | 3 | 1
Dysgeusia (Nervous system disorders) | 3 | 2 | 0
Tremor (Nervous system disorders) | 2 | 1 | 0
Memory impairment (Nervous system disorders) | 2 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 0 | 0
Paraesthesia (Nervous system disorders) | 2 | 0 | 0
Amnesia (Nervous system disorders) | 1 | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 2 | 0
Thrombosis in device (Product Issues) | 2 | 3 | 0
Insomnia (Psychiatric disorders) | 8 | 4 | 0
Anxiety (Psychiatric disorders) | 4 | 2 | 0
Depression (Psychiatric disorders) | 3 | 1 | 0
Delirium (Psychiatric disorders) | 1 | 2 | 0
Confusional state (Psychiatric disorders) | 0 | 2 | 0
Hallucination (Psychiatric disorders) | 2 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 3 | 0
Haematuria (Renal and urinary disorders) | 2 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 2 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 2 | 0
Nocturia (Renal and urinary disorders) | 2 | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 3 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 4 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 3 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 3 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Hypotension (Vascular disorders) | 2 | 6 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 1 | 0
Hypertension (Vascular disorders) | 3 | 0 | 0
Phlebitis (Vascular disorders) | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.